CLINICAL TRIAL: NCT02996552
Title: Annuloplasty for the Treatment of Not-Severe Tricuspid Regurgitation in Patients Undergoing Surgery for Mitral Valve Disease: a Prospective, Spontaneous, Multicentre, Randomized Study
Brief Title: Annuloplasty for Not-Severe TR in Patients Undergoing MV Repair Versus Mitral Repair Only (NOSTRUM)
Acronym: NOSTRUM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale San Raffaele (Other)
Collaborators: Istituto Clinico Humanitas (Other); Central Clinical Hospital of the Ministry of Internal Affairs and Administration, Warsaw, Poland (Other)
Responsible Party: Principal Investigator, Michele De Bonis, Associate Professor, Ospedale San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 072/11
Record Dates: First submitted 2016-12-06; First posted 2016-12-19 (Estimated); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Tricuspid Disease; Mitral Regurgitation
Keywords: Tricuspid annulus dilation; mitral valve regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- M & T Repair Group (Experimental): Both mitral and tricuspid valves repair
  Interventions: Procedure: M & T Repair Group
- Mitral-Only Group (Active Comparator): Only mitral valve repair
  Interventions: Procedure: Mitral-Only Group

INTERVENTIONS:
Procedure: M & T Repair Group — After the mitral valve repair a device for tricuspid annuloplasty will be implanted.
  Arms: M & T Repair Group
Procedure: Mitral-Only Group — Mitral valve repair alone; after the mitral valve repair no device for tricuspid annuloplasty will be implanted.
  Arms: Mitral-Only Group

SUMMARY:
The surgical treatment of less than severe (≤2+/4+) functional tricuspid regurgitation (TR) in patient undergoing mitral valve surgery, is still controversial: some observational studies have suggested that performing tricuspid annuloplasty in patients undergoing mitral valve surgery with a dilated tricuspid annulus, and TR≤2+ may provide a clinical benefit, while in other observational studies such benefit has not been documented.

The ESC Guidelines assign the class IIa recommendation for surgical treatment in patients with tricuspid regurgitation ≤2+ and a dilated annulus, if surgery is concomitant to the repair or replacement of the mitral valve. However the level of evidence C (expert opinion) confirms the absence of clear scientific evidence to support this recommendation.

It is therefore very important to carry out randomized trials designed to really prove the supposed efficacy of prophylactic tricuspid annuloplasty, especially in patients with degenerative etiology where the data are particularly controversial.

The aim of the study will be to establish the effectiveness of the tricuspid annuloplasty in the early stage of TR. The investigators enrolled patients with TR≤2+ and annular dilation undergoing mitral valve repair.

Primary end-point will be the freedom from recurrence of TR≥3+ and from progression of 2 degrees of TR compared to pre-operative, at discharge and 12 months after surgery, assessment by transthoracic echocardiography. Secondary endpoints are to demonstrate the superiority of combined treatment (M & T Repair Group) compared to single treatment (Mitral-Only Group) at 5 and 10 years after surgery.

This will be an experimental superiority, prospective, spontaneous, multicenter, randomized trial.

Patients will be randomly assigned to two parallel arms with an allocation ratio 1:1 stratified by center, to receive mitral repair only (Mitral-Only group) or both mitral and tricuspid repair (M & T Repair group).

DETAILED DESCRIPTION:
Current guidelines recommend surgical treatment of secondary tricuspid regurgitation (TR) in patients with mild or moderate TR undergoing mitral valve (MV) surgery if significant dilatation of the tricuspid annulus is documented. Indeed, several observational series and small randomized studies have shown that in the presence of tricuspid annulus dilatation, not treating less than severe secondary TR may lead to progression of the tricuspid disease despite correction of the associated left-sided lesion.

However, the level of evidence C (expert opinion) confirms the absence of clear scientific evidence to support this recommendation.

It is therefore very important to carry out randomized trials designed to really prove the supposed efficacy of prophylactic tricuspid annuloplasty, especially in patients with degenerative etiology where the data are particularly controversial.

The aim of the study will be to establish the effectiveness of the tricuspid annuloplasty in the early stage. The investigators enrolled patient with TR≤2+ and annular dilation undergoing mitral valve repair.

This will be a multicenter single-blind parallel group randomized controlled trial. Patients will be randomly assigned to two parallel arms with an allocation ratio 1:1, to receive one of two surgical procedures. Patients that will match the inclusion criteria at the preoperative evaluation will be recruited.

Patient will be randomized according to a computer-generated list of casual numbers. Information about patient allocation will be kept in closed opaque envelopes and nobody will know patient allocation before randomization. Patients will be blind to allocation.

The day of surgery patients will be subsequently randomized into two arms with an allocation ratio 1:1 stratified by center, to receive:

1. M & T Repair Group
2. Mitral-Only Group Each group will consist of 71 patients. All patients will receive the mitral valve repair and in patients enrolled in the M & T Repair Group an Edwards MC3 Tricuspid ring will be implanted.

Primary end-point will be the freedom from recurrence of TR≥3+ and from progression of 2 degrees of TR compared to pre-operative, at discharge and 12 months after surgery, assessment by transthoracic echocardiography. Secondary endpoints are to demonstrate the superiority of combined treatment (M & T Repair Group) compared to single treatment (Mitral-Only Group) at 5 and 10 years after surgery.

For statistical analysis the data will be expressed as "average ± standard deviation" or as percentage. A "probability value" less than 0.05 will be considered as "statistically significant." Outcomes will be compared using the "X2" analysis for categorical variables and the "t-test" for the continuous onces. The data will be analyzed using SPSS version 11.5 (SPSS Inc., Chicago, IL, USA) for Windows (Microsoft Corp, Redmond, WA). Survival and freedom from reoperation, freedom from TR≥3+ or from a progression of TR of at least 2 grades (as compared to baseline), will be analyzed by the method of Kaplan-Meier. The analysis "univariate" and possibly "multivariate" of risk factors will be performed with "Cox proportional hazards regression".

The Fine and Gray model will be used in a "competing risk analysis" for "time to TR ≥ 3+/4+" and "time to TR progression of at least 2 grades compared to baseline" considering the death event as competitive risk.

In addition, estimates of the respective cumulative incidence (CIF) of these events in the 2 groups will be compared to determine the impact on such endpoints of the execution or non-execution of tricuspid anuloplasty.

The aim of the study is to demonstrate the superiority of combined mitral and tricuspid treatment (M & T Repair) compared to isolated mitral repair (Mitral-Only Group) in the enrolled patients.

The primary end-point is to demonstrate that, at 1 year of follow-up, the recurrence of TR≥3+ or the progression of TR of at least 2 degrees (compared to baseline) occurs in less than 1% of the patients undergoing both mitral e tricuspid repair (M & T Repair Group). The expected rate for the Mitral-Only group is 15%. (Power = 80%, alpha = 0.05, Number of Patients per group = 71).

Secondary endpoints are to demonstrate the superiority of the combined treatment (M & T Repair Group) compared to the single treatment (Mitral-Only Group) at 5 and 10 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years;
* ability to provide informed consent;
* patients scheduled for mitral valve regurgitation
* TR ≤ 2+ with annular dilation
* Tricuspid diastolic diameter ≥ 40 mm or 21 mm/m2

Exclusion Criteria:

* patient's refusal
* non-elective cardiac surgery;
* organic disease of tricuspid valve
* TR≥3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2011-06-08 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
The 1-year freedom from recurrence of TR≥3+ and from progression by 2 degrees compared to pre-operative. | 1 year

SECONDARY OUTCOMES:
The 5-year freedom from recurrence of TR >= 3+ and from progression by 2 degrees compared to pre-operative, in the combined treatment group (M & T Repair Group) and in the single treatment group ( Mitral-Only Group) | 5 years
The 10-year freedom from recurrence of TR >= 3+ and from progression by 2 degrees compared to pre-operative, in the combined treatment group (M & T Repair Group) and in the single treatment group ( Mitral-Only Group) | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Michele De Bonis, MD,FESC,FAHA, Principal Investigator — IRCCS Ospedale San Raffale Milano
Locations (3):
- Italy (2):
  - Istituto Clinico Humanitas, Rozzano, Milano
  - IRCCS Ospedale San Raffaele, Milan
- Central Clinical Hospital of the Ministry of Internal Affairs and Administration, Warsaw, Poland, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No